CLINICAL TRIAL: NCT01190878
Title: A Randomized Double-masked 14-day Study to Compare the Ocular Safety, Tolerability, and Efficacy of Differing Dosing Regimens of ISV-303 to Vehicle and Xibrom™ in Post Cataract Surgery Volunteers
Brief Title: Study to Compare Differing Dosing Regimens of ISV-303 (Bromfenac in DuraSite) to Xibrom and Vehicle in Post Cataract Surgery Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-10-303-001
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Ocular Inflammation
MeSH Terms: interventions — bromfenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ISV-303 BID (Experimental)
  Interventions: Drug: ISV-303
- ISV-303 QD (Experimental)
  Interventions: Drug: ISV-303
- Xibrom BID (Active Comparator)
  Interventions: Drug: Xibrom™
- DuraSite Vehicle BID (Placebo Comparator)
  Interventions: Drug: DuraSite Vehicle

INTERVENTIONS:
Drug: ISV-303 — 0.075% of bromfenac in DuraSite dosed QD
  Arms: ISV-303 QD
Drug: ISV-303 — 0.075% of bromfenac in DuraSite dosed BID
  Arms: ISV-303 BID
Drug: DuraSite Vehicle — Vehicle dosed BID
  Arms: DuraSite Vehicle BID
Drug: Xibrom™ — 0.09% bromfenac dosed BID
  Arms: Xibrom BID

SUMMARY:
The purpose of this study is to evaluate the ocular safety, tolerability, and efficacy in topical administration of differing dosing regimens of ISV-303 compared to vehicle and Xibrom™ when dosed for 2 weeks in post-cataract-surgery volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral cataract surgery (phacoemulsification or extracapsular extraction) with posterior chamber intraocular lens implantation on the day prior to study enrollment
* Meet the best corrected visual acuity score requirement
* Meet the IOP requirement
* Additional inclusion criteria also apply

Exclusion Criteria:

* Known hypersensitivity or poor tolerance to bromfenac sodium or any component of the study medications or any of the procedural medications
* Use of any ocular topical, or systemic medication that could interfere with normal lacrimation, wound healing, the test agent, or the interpretation of study results, within 1 week prior to Day of Surgery
* Additional exclusion criteria also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

REFERENCES:
- [Derived] Trattler W, Hosseini K. Twice-Daily vs. Once-Daily Dosing with 0.075% Bromfenac in DuraSite: Outcomes from a 14-Day Phase 2 Study. Ophthalmol Ther. 2017 Dec;6(2):277-284. doi: 10.1007/s40123-017-0102-x. Epub 2017 Aug 17. PMID 28819932

RESULTS

PARTICIPANT FLOW:
Groups:
- ISV-303 BID: ISV-303: 0.075% bromfenac in DuraSite dosed BID
- ISV-303 QD: ISV-303: 0.075% bromfenac in DuraSite dosed QD
Period: Overall Study
Arm/Group | ISV-303 BID | ISV-303 QD | Xibrom BID | DuraSite Vehicle BID
Started | 40 | 45 | 42 | 42
Completed | 37 | 42 | 37 | 22
Not Completed | 3 | 3 | 5 | 20

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Xibrom BID: Xibrom™: Xibrom dosed BID
- Total: Total of all reporting groups
Arm/Group | ISV-303 BID | ISV-303 QD | Xibrom BID | DuraSite Vehicle BID | Total
Number analyzed (Participants) | 40 | 45 | 42 | 42 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (7.70) | 70.9 (9.75) | 68.6 (10.49) | 67.0 (9.30) | 69.5 (9.47)
Age, Customized [Number; unit: participants]
  18-30 years | 0 | 0 | 1 | 0 | 1
  31-50 years | 0 | 0 | 0 | 2 | 2
  51-70 years | 22 | 22 | 22 | 25 | 91
  >70 years | 18 | 23 | 19 | 15 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 20 | 24 | 89
  Male | 16 | 24 | 22 | 18 | 80

OUTCOME MEASURES:

1. Primary Outcome: Ocular Inflammation
Description: Anterior Chamber Cell Grade 0 at Day 15 measured on a 0 to 4 scale: "0" is 0 cells; "1" is 1-10 cells; "2" is 11-20 cells; "3" is 21-50 cells; "4" is > 50 cells.
Time Frame: 15 days
Population: Intent-to-Treat (ITT) Population using Last Observation Carried Forward (LOCF) method.
Measure: Number; unit: participants
Arm/Group | ISV-303 BID | ISV-303 QD | Xibrom BID | DuraSite Vehicle BID
Number analyzed (Participants) | 40 | 45 | 42 | 42
participants | 21 | 24 | 18 | 8

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | ISV-303 BID | ISV-303 QD | Xibrom BID | DuraSite Vehicle BID
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/45 | 1/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 4/45 | 1/42 | 1/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-303 BID (N=40) | ISV-303 QD (N=45) | Xibrom BID (N=42) | DuraSite Vehicle BID (N=42)
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-303 BID (N=40) | ISV-303 QD (N=45) | Xibrom BID (N=42) | DuraSite Vehicle BID (N=42)
Iritis (Eye disorders) | 0 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other